CLINICAL TRIAL: NCT04140266
Title: Phase 3B, Randomized, Open-Label, Safety, and Drug Detection Study of Dapivirine Vaginal Ring and Oral TRUVADA® in Breastfeeding Mother-Infant Pairs
Brief Title: Safety and Drug Detection Study of Dapivirine Vaginal Ring and Oral TRUVADA® in Breastfeeding Mother-Infant Pairs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTN-043; 38591 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Contraceptive Devices, Female; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 (Experimental): Mothers will use one DPV VR continuously for approximately one month, replacing the DPV VR each month for approximately three months.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)-004
- Group B: Truvada Tablet (Experimental): Mothers will take one Truvada oral tablet daily for approximately three months.
  Interventions: Drug: Truvada Tablet

INTERVENTIONS:
Drug: Dapivirine (DPV) Vaginal Ring (VR)-004 — Vaginal ring containing 25 mg of DPV
  Arms: Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Drug: Truvada Tablet — Oral tablet containing 200 mg emtricitabine (FTC)/300 mg tenofovir disoproxil fumarate (TDF)
  Other Names: Emtricitabine/Tenofovir Disoproxil Fumarate; FTC/TDF
  Arms: Group B: Truvada Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and drug detection of the dapivirine vaginal ring and oral Truvada in breastfeeding mother-infant pairs.

DETAILED DESCRIPTION:
This study will evaluate the safety and drug detection of the dapivirine (DPV) vaginal ring (VR) and oral Truvada in breastfeeding mother-infant pairs.

Mother-infant pairs will be randomly assigned to receive either the DPV VR or oral Truvada. Mothers randomized to the DPV VR will use the VR continuously for approximately one month (4 weeks), replacing the VR each month for approximately three months (12 weeks). Mothers using the Truvada tablet will take one tablet by mouth daily for approximately three months (12 weeks).

Study visits will occur at Day 0, Weeks 1 and 2, and Months 1, 2, 3, and 3.5. Study visits may include behavioral assessments; product acceptability assessments; infant feeding assessments; physical examinations; blood, urine, and breast milk collection; and pelvic examination and specimen collection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Mother

Participant mothers must meet all the following criteria to be eligible for inclusion in the study:

* Age 18 years or older at Screening, as verified per site Standard Operating Procedures (SOPs).
* At Enrollment, between 6 to 12 weeks postpartum (verified by birth records and/or similar supportive documentation and defined as between 42 - 84 days after delivery, inclusive).
* By participant report at Screening and Enrollment, currently exclusively breastfeeding one infant and willing and able to continue exclusively breastfeeding that infant for the duration of their participation in the study.

  * Note: Exclusive breastfeeding will be defined as infant nutrition solely from breast milk, as determined by 7-day recall breastfeeding history. For the purposes of MTN-043, "breastfeeding" refers to all human milk feeding situations when an infant is fed with participant's own human milk whether the milk is received directly from the breast or as expressed milk.
* Consistently using an effective method of contraception per participant report at Enrollment, and intending to continue use of an effective method for the duration of study participation. Effective methods include contraceptive implants, intrauterine device, injectable progestin, oral contraceptive pills, and surgical sterilization.
* Able and willing to comply with all study requirements and complete all study procedures.
* Able and willing to provide the following:

  * Written informed consent to be screened for and to take part in the study.
  * Written informed consent for the breastfed infant to be screened for and take part in the study.
* Intention to stay within study catchment area for study duration and willingness to give adequate locator information, as defined in site SOPs.
* At Screening and Enrollment, HIV-uninfected based on HIV testing performed by study staff (per algorithm in the study protocol).
* At Screening and Enrollment, willing to be randomized at time of enrollment to either of the study products, and to continue study product use for at least 12 weeks.

Inclusion Criteria - Infant

Each mother eligible for MTN-043 will be asked to provide written informed consent for herself and her infant to participate in the study if the infant meets the following criteria:

* At Screening and Enrollment, infant is exclusively breastfed.

  * Note: Exclusive breastfeeding will be defined as infant nutrition solely from breast milk, as determined by 7-day recall breastfeeding history. For the purposes of MTN-043, "breastfeeding" refers to all human milk feeding situations when an infant is fed with participant's own human milk whether the milk is received directly from the breast or as expressed milk.
* At Screening and Enrollment, the infant is generally healthy, according to the judgment of the investigator of record (IoR)/designee.
* At Enrollment, the infant is between the ages of 6 and 12 weeks postpartum (verified by birth records and/or similar supportive documentation with age defined as between 42 - 84 days after delivery, inclusive).

Exclusion Criteria:

Exclusion Criteria - Mother

Mothers who meet any of the following criteria will be excluded from the study:

* At Screening or Enrollment, breastfeeding infant ineligible for enrollment in the study.
* At Screening or Enrollment, participant reports any of the following:

  * Known adverse reaction to any of the study products (ever).
  * Known adverse reaction to latex and polyurethane (ever).
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to Enrollment.
  * Use of vaginal medications(s) or other vaginal products within five days prior to Enrollment.
  * Non-therapeutic injection drug use in the 12 months prior to Enrollment.
  * History of exposure to any investigational drug(s) during pregnancy, including participation in MTN-042.
* At Screening or Enrollment, has a positive HIV test.
* At Screening or Enrollment, Grade 2 or higher breast or genitourinary findings.
* At Screening or Enrollment, has a positive urinary pregnancy test.
* At Screening, has any of the following laboratory abnormalities:

  * Positive for hepatitis B surface antigen (HBsAg).
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≥ Grade 2.
  * Creatinine ≥ Grade 1.
  * Estimated creatinine clearance ≥ Grade 2 (Cockcroft Gault formula).
* Diagnosed with urinary tract infection (UTI), pelvic inflammatory disease (PID), sexually transmitted infection (STI) or reproductive tract infection (RTI), requiring treatment per World Health Organization (WHO) Guidelines.

  * Note: Otherwise eligible participants diagnosed during Screening with a UTI, PID or STI/RTI requiring treatment per WHO Guidelines - other than asymptomatic bacterial vaginosis (BV) and asymptomatic vulvovaginal candidiasis - are offered treatment consistent with WHO recommendations and may be enrolled after completing treatment if all symptoms have resolved. If treatment is completed and symptoms have resolved prior to obtaining informed consent for Screening, the participant may be enrolled. Genital warts requiring treatment also must be treated prior to enrollment. Genital warts requiring treatment are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
* As determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* At Enrollment, participant reports any of the following:

  * Participation in any research study involving drugs, vaccines, or medical devices 30 days or less prior to enrollment.
  * Currently participating in other research studies involving drugs, vaccines, or medical devices.
  * Expected to participate in other research studies involving drugs, vaccines, or medical devices during study participation.

Exclusion Criteria - Infants

* Has any condition that, in the opinion of the IoR/designee, would preclude eligibility, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

  * Note: Examples of exclusionary infant conditions include clinical evidence of stunting or illness.
* At Enrollment, according to the report of the mother, any of the following apply for the infant:

  * Infants with birth weight less than 2000g.
  * Participation in any research study involving drugs, vaccines, or medical devices since birth.
  * Currently participating in other research studies involving drugs, vaccines, or medical devices.
  * Expected to participate in other research studies involving drugs, vaccines, or medical devices for the duration of study participation.

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxensia Owor, MBChB, MMed, MPH, Study Chair — MU-JHU CARE; Lisa Noguchi, PhD, CNM, Study Chair — Johns Hopkins Bloomberg School of Public Health; Jen Balkus, PhD, MPH, Study Chair — Hans Rosling Center for Population Health
Locations (4):
- Blantyre CRS (Johns Hopkins Research Project/College of Medicine), Blantyre, Malawi
- Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng, South Africa
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Zengeza CRS, Chitungwiza, Mashonaland East Province, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to researchers upon request. The IPD to be shared will be negotiated with the researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 8 weeks of request approval and to be available as long as needed.
Access Criteria: MTN-043 study management team approval

REFERENCES:
- [Derived] Noguchi LM, Owor M, Mgodi NM, Gati Mirembe B, Dadabhai S, Horne E, Gundacker H, Richardson BA, Bunge K, Scheckter R, Song M, Marzinke MA, Anderson PL, Livant E, Jacobson C, Piper JM, Chakhtoura N, Hillier SL, Balkus JE; MTN-043 Study Team. Safety and drug quantification of the dapivirine vaginal ring and oral pre-exposure prophylaxis in breastfeeding mother-infant pairs (MTN-043): a phase 3B, open-label, randomised trial. Lancet HIV. 2025 Mar;12(3):e180-e190. doi: 10.1016/S2352-3018(24)00306-0. Epub 2025 Feb 12. PMID 39954697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 197 mother-infant pairs were enrolled in 4 African countries from September 2020 until July 2021.
Pre-assignment Details: 197 mother-infant pairs were enrolled in the study. When the mothers are enrolled and discontinued from the study, their infants are enrolled or discontinued.
Period: Overall Study
Arm/Group | Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Group B: Truvada Tablet
Started (Mothers and infants are added as two milestones.) | 296 | 98
Mothers | 148 | 49
Infants | 148 | 49
Completed | 290 | 96
Not Completed | 6 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Adverse Events for Mothers randomized to the DPV VR study arm.
- Mothers - Group B: Truvada Tablet: Adverse Events for Mothers randomized to the Truvada oral tablet study arm.
- Infants - Group A: DPV VR: Adverse Events for Infants of Mothers randomized to the DPV VR study arm.
- Infants - Group B: Truvada Tablet: Adverse Events for Infants of Mothers randomized to the Truvada oral tablet study arm.
- Total: Total of all reporting groups
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet | Infants - Group A: DPV VR | Infants - Group B: Truvada Tablet | Total
Number analyzed (Participants) | 148 | 49 | 148 | 49 | 394
Age, Continuous [Median (Full Range); unit: years] — Population: Only mothers are included in this baseline measure since mother age is summarized in years. Infants age is summarized below in weeks.
  years
    Mothers' Age, years: number analyzed (Participants) | 148 | 49 | 0 | 0 | 197
    Mothers' Age, years | 26 [18 to 43] | 25 [18 to 38] |  |  | 26 [18 to 43]
Age, Continuous [Median (Full Range); unit: weeks] — Population: Only infants are included in this baseline measure since infant age is summarized in weeks.
  weeks
    Infants' Age, weeks: number analyzed (Participants) | 0 | 0 | 148 | 49 | 197
    Infants' Age, weeks |  |  | 9 [6 to 12] | 8 [6 to 12] | 9 [6 to 12]
Age, Customized [Count of Participants; unit: Participants] — Population: Only mothers are included in this baseline measure since mothers age is in years. Infants are categorized below in weeks.
  Participants
    mother age: number analyzed (Participants) | 148 | 49 | 0 | 0 | 197
    mother age: 18-19 years | 14 | 5 | 0 | 0 | 19
    mother age: 20-24 years | 50 | 17 | 0 | 0 | 67
    mother age: 25-29 years | 42 | 12 | 0 | 0 | 54
    mother age: 30-34 years | 28 | 12 | 0 | 0 | 40
    mother age: 35-39 years | 13 | 3 | 0 | 0 | 16
    mother age: 40-45 years | 1 | 0 | 0 | 0 | 1
Age, Customized [Count of Participants; unit: Participants] — Population: Only infants are included in this baseline measure since infant age is categorized in weeks.
  Participants
    Infant age: number analyzed (Participants) | 0 | 0 | 148 | 49 | 197
    Infant age: 6 to 9 weeks | 0 | 0 | 87 | 34 | 121
    Infant age: >9 weeks to 12 weeks | 0 | 0 | 61 | 15 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 49 | 84 | 24 | 305
  Male | 0 | 0 | 64 | 25 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 148 | 49 | 148 | 49 | 394
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 148 | 49 | 148 | 49 | 394
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 29 | 10 | 29 | 10 | 78
  South Africa | 27 | 9 | 27 | 9 | 72
  Uganda | 42 | 13 | 42 | 13 | 110
  Zimbabwe | 50 | 17 | 50 | 17 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Mother Participants With Serious Adverse Events (SAEs) Including Maternal Deaths in Both Study Arms
Description: As defined by the Manual for Expedited Reporting of Adverse Events to the Division of AIDS (DAIDS) (Version 2.0, January 2010)
Time Frame: Measured through Month 3.5
Population: All Mothers received study product and are used in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 148 | 49
Participants | 2 | 0

2. Primary Outcome: Number of Mother Participants With Grade 3 or Higher Adverse Events (AEs) in Both Study Arms
Description: As defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])
Time Frame: Measured through Month 3.5
Population: All enrolled mothers received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Group B: Truvada Tablet
Number analyzed (Participants) | 148 | 49
Participants | 3 | 2

3. Primary Outcome: Number of Infant Participants With SAEs Including Infant Deaths in Both Study Arms
Description: As defined by the Manual for Expedited Reporting of Adverse Events to DAIDS (Version 2.0, January 2010)
Time Frame: Measured through Month 3.5
Population: All infants were exposed to study product through mothers' breastmilk. All enrolled mothers received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Infants - Group A: DPV VR | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 148 | 49
Participants | 4 | 0

4. Primary Outcome: Number of Infant Participants With Grade 3 or Higher AEs in Both Study Arms
Description: As defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Time Frame: Measured through Month 3.5
Population: Infants were exposed to study product through breastmilk. All enrolled mothers received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Infants - Group A: DPV VR | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 148 | 49
Participants | 10 | 1

5. Primary Outcome: Number and Proportion of Mothers With Detectable Plasma Dapivirine (DPV) Concentrations
Description: This endpoint is based on DPV concentration laboratory results from evaluable plasma specimens from mother participants. DPV concentrations above the lower limit of quantification (LLOQ) are considered detectable. For DPV concentration in plasma, the LLOQ is 20 pg/ml. The infant endpoint is included as a separate section below.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the DPV VR arm with available and evaluable plasma specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infant results are in a separate section below.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Mothers randomized to the DPV Vaginal Ring study arm with evaluable plasma specimens.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Number analyzed (Participants) | 147
Participants
  Week 1: number analyzed (Participants) | 140
  Week 1 | 139
  Week 2: number analyzed (Participants) | 140
  Week 2 | 136
  Month 1: number analyzed (Participants) | 141
  Month 1 | 139
  Month 2: number analyzed (Participants) | 144
  Month 2 | 138
  Product Use End Visit: number analyzed (Participants) | 139
  Product Use End Visit | 136
  Study End Visit: number analyzed (Participants) | 142
  Study End Visit | 48

6. Primary Outcome: Number and Proportion of Mothers With Detectable Emtricitabine Triphosphate (FTC-TP) Concentrations
Description: This endpoint is based on FTC-TP concentration laboratory results from evaluable dried blood spot (DBS) specimens from mother participants. FTC-TP concentrations above the lower limit of quantification (LLOQ) are considered detectable. For FTC-TP concentration in DBS specimens, the LLOQ is 0.125 pmol/punch. The infant endpoint is included as a separate section below.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the Truvada arm with available and evaluable DBS specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infant results are in a separate section below.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group B: Truvada Tablet: Mothers randomized to the Truvada oral tablet study arm with evaluable Dried Blood Spot specimens,
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 1: number analyzed (Participants) | 47
  Week 1 | 45
  Week 2 | 46
  Month 1: number analyzed (Participants) | 47
  Month 1 | 38
  Month 2: number analyzed (Participants) | 44
  Month 2 | 34
  Product Use End Visit: number analyzed (Participants) | 47
  Product Use End Visit | 38
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 1

7. Primary Outcome: Number and Proportion of Mothers With Detectable Tenofovir Diphosphate (TFV-DP) Concentrations
Description: This endpoint is based on TFV-DP concentration laboratory results from evaluable dried blood spot (DBS) specimens from mother participants. TFV-DP concentrations above the lower limit of quantification (LLOQ) are considered detectable. For TFV-DP concentrations, the LLOQ is 31.3 fmol/punch. The infant endpoint is included as a separate section below.
Time Frame: Measured through Month 3.5
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 1: number analyzed (Participants) | 47
  Week 1 | 47
  Week 2 | 48
  Month 1: number analyzed (Participants) | 47
  Month 1 | 45
  Month 2: number analyzed (Participants) | 44
  Month 2 | 44
  Product Use End Visit: number analyzed (Participants) | 47
  Product Use End Visit | 47
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 45

8. Primary Outcome: Number and Proportion of Mothers With Detectable Breastmilk DPV Concentrations
Description: This endpoint is based on DPV concentration laboratory results from evaluable breastmilk specimens from mother participants. DPV concentrations above the lower limit of quantification (LLOQ) are considered detectable. For DPV concentration in breastmilk, the LLOQ is 10 pg/ml.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the DPV VR arm with available and evaluable breastmilk specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infants are not included in this population.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Mothers randomized to the DPV Vaginal Ring study arm with evaluable breast milk specimens.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Number analyzed (Participants) | 146
Participants
  Week 1: number analyzed (Participants) | 138
  Week 1 | 137
  Week 2: number analyzed (Participants) | 139
  Week 2 | 137
  Month 1: number analyzed (Participants) | 140
  Month 1 | 138
  Month 2: number analyzed (Participants) | 142
  Month 2 | 138
  Product Use End Visit: number analyzed (Participants) | 138
  Product Use End Visit | 135
  Study End Visit: number analyzed (Participants) | 142
  Study End Visit | 94

9. Primary Outcome: Number and Proportion of Mothers With Detectable Breastmilk FTC Concentrations
Description: This endpoint is based on FTC concentration laboratory results from evaluable breastmilk specimens from mother participants. FTC concentrations above the lower limit of quantification (LLOQ) are considered detectable. For FTC concentrations in breastmilk, the LLOQ is 5 mg/ml.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the Truvada arm with available and evaluable breastmilk specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infants are not included in this population.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group B: Truvada Tablet: Mothers randomized to the Truvada oral tablet study arm with evaluable breast milk specimens,
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 1 | 47
  Week 2: number analyzed (Participants) | 47
  Week 2 | 45
  Month 1: number analyzed (Participants) | 47
  Month 1 | 44
  Month 2: number analyzed (Participants) | 43
  Month 2 | 39
  Product Use End Visit: number analyzed (Participants) | 46
  Product Use End Visit | 40
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 1

10. Primary Outcome: Number and Proportion of Mothers With Detectable Breastmilk TFV Concentrations
Description: This endpoint is based on TFV concentration laboratory results from evaluable breastmilk specimens from mother participants. TFV concentrations above the lower limit of quantification (LLOQ) are considered detectable. For TFV concentrations in breastmilk, the LLOQ is 1 ng/ml.
Time Frame: Measured through Month 3.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 1 | 47
  Week 2: number analyzed (Participants) | 47
  Week 2 | 44
  Month 1: number analyzed (Participants) | 47
  Month 1 | 42
  Month 2: number analyzed (Participants) | 43
  Month 2 | 38
  Product Use End Visit: number analyzed (Participants) | 46
  Product Use End Visit | 38
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 3

11. Primary Outcome: Number and Proportion of Infants With Detectable Plasma DPV Concentrations
Description: This endpoint is based on DPV concentration laboratory results from evaluable plasma specimens from infant participants. DPV concentrations above the lower limit of quantification (LLOQ) are considered detectable. For DPV concentration in plasma, the LLOQ is 20 pg/ml. The mother endpoints are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the infants of mothers randomized to the DPV VR arm with available and evaluable plasma specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes infants with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Mother results are in a separate section above.
Measure: Count of Participants; unit: Participants
Groups:
- Infants - Group A: DPV VR: Infants of Mothers randomized to the DPV VR study arm.
Arm/Group | Infants - Group A: DPV VR
Number analyzed (Participants) | 147
Participants
  Week 2: number analyzed (Participants) | 140
  Week 2 | 21
  Month 1: number analyzed (Participants) | 139
  Month 1 | 20
  Month 2: number analyzed (Participants) | 143
  Month 2 | 14
  Product Use End Visit: number analyzed (Participants) | 138
  Product Use End Visit | 7
  Study Exit Visit: number analyzed (Participants) | 142
  Study Exit Visit | 0

12. Primary Outcome: Number and Proportion of Infants With Detectable FTC-TP Concentrations
Description: This endpoint is based on FTC-TP concentration laboratory results from evaluable dried blood spot (DBS) specimens from infant participants. FTC-TP concentrations above the lower limit of quantification (LLOQ) are considered detectable. For FTC-TP concentrations from DBS specimens, the LLOQ is 0.125 pmol/punch. The mother endpoints are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the infants of mothers randomized to the Truvada arm with available and evaluable DBS specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes infants with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Mother results are in a separate section above.
Measure: Count of Participants; unit: Participants
Groups:
- Infants - Group B: Truvada Tablet: Infants of Mothers randomized to the Truvada oral tablet study arm.
Arm/Group | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 2: number analyzed (Participants) | 47
  Week 2 | 4
  Month 1: number analyzed (Participants) | 47
  Month 1 | 2
  Month 2: number analyzed (Participants) | 45
  Month 2 | 2
  Product Use End Visit: number analyzed (Participants) | 45
  Product Use End Visit | 1
  Study Exit Visit: number analyzed (Participants) | 46
  Study Exit Visit | 0

13. Primary Outcome: Number and Proportion of Infants With Detectable TFV-DP Concentrations
Description: This endpoint is based on TFV-DP concentration laboratory results from evaluable dried blood spot (DBS) specimens from infant participants. TFV-DP concentrations above the lower limit of quantification (LLOQ) are considered detectable. For TFV-DP concentrations from DBS specimens, the LLOQ is 31.3 fmol/punch. The mother endpoints are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 48
Participants
  Week 2: number analyzed (Participants) | 47
  Week 2 | 0
  Month 1: number analyzed (Participants) | 47
  Month 1 | 0
  Month 2: number analyzed (Participants) | 45
  Month 2 | 0
  Product Use End Visit: number analyzed (Participants) | 45
  Product Use End Visit | 0
  Study Exit Visit: number analyzed (Participants) | 46
  Study Exit Visit | 0

14. Primary Outcome: Geometric Mean of Maternal DPV Concentrations From Plasma by Visit
Description: This endpoint is based on DPV concentration laboratory results from evaluable plasma specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the DPV VR arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (20pg/ml). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Number analyzed (Participants) | 147
pg/mL
  Week 1: number analyzed (Participants) | 140
  Week 1 | 327.9 (61.3)
  Week 2: number analyzed (Participants) | 140
  Week 2 | 314.9 (92.1)
  Month 1: number analyzed (Participants) | 141
  Month 1 | 275.4 (76.9)
  Month 2: number analyzed (Participants) | 144
  Month 2 | 263.8 (111.9)
  Product Use End Visit: number analyzed (Participants) | 139
  Product Use End Visit | 260.4 (87.3)
  Study End Visit: number analyzed (Participants) | 142
  Study End Visit | 16.7 (93.5)

15. Primary Outcome: Geometric Mean of Maternal FTC-TP Concentrations by Visit
Description: This endpoint is based on FTC-TP concentration laboratory results from evaluable dried blood spot (DBS) specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (0.125 pmol/punch). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/punch
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
pmol/punch
  Week 1: number analyzed (Participants) | 47
  Week 1 | 0.3 (51.3)
  Week 2 | 0.3 (58.4)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 0.3 (91.5)
  Month 2: number analyzed (Participants) | 44
  Month 2 | 0.2 (90.9)
  Product Use End Visit: number analyzed (Participants) | 47
  Product Use End Visit | 0.2 (91.3)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 0.1 (21.9)

16. Primary Outcome: Geometric Mean of Maternal TFV-DP Concentrations by Visit
Description: This endpoint is based on TFV-DP concentration laboratory results from evaluable dried blood spot (DBS) specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (31.3 fmol/punch). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/punch
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
fmol/punch
  Week 1: number analyzed (Participants) | 47
  Week 1 | 254.6 (62.8)
  Week 2 | 424.2 (65.2)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 524.7 (117.8)
  Month 2: number analyzed (Participants) | 44
  Month 2 | 551.9 (97.5)
  Product Use End Visit: number analyzed (Participants) | 47
  Product Use End Visit | 591.5 (135.5)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 330.8 (137.8)

17. Primary Outcome: Geometric Mean of Maternal DPV Concentrations From Breastmilk by Visit
Description: This endpoint is based on DPV concentration laboratory results from evaluable breastmilk specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the DPV VR arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (10pg/ml). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the DPV VR arm with available and evaluable breastmilk specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infant results are in a separate section below.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Number analyzed (Participants) | 146
pg/mL
  Week 1: number analyzed (Participants) | 138
  Week 1 | 529.4 (108.0)
  Week 2: number analyzed (Participants) | 139
  Week 2 | 492.0 (122.3)
  Month 1: number analyzed (Participants) | 140
  Month 1 | 457.0 (119.3)
  Month 2: number analyzed (Participants) | 142
  Month 2 | 418.9 (545.0)
  Product Use End Visit: number analyzed (Participants) | 138
  Product Use End Visit | 402.8 (154.5)
  Study End Visit: number analyzed (Participants) | 142
  Study End Visit | 20.0 (210.7)

18. Primary Outcome: Geometric Mean of Maternal FTC Concentrations From Breastmilk by Visit
Description: This endpoint is based on FTC concentration laboratory results from evaluable breastmilk specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (5 mg/ml). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: This endpoint includes the mothers randomized to the Truvada arm with available and evaluable breastmilk specimens at the specific timepoint. The "Overall Number of Participants Analyzed" includes mothers with an evaluable specimen for at least one timepoint. Evaluable is defined as the specimens that were successfully tested at the central laboratory. Infant results are in a separate section below.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mL
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
mg/mL
  Week 1 | 552.6 (167.4)
  Week 2: number analyzed (Participants) | 47
  Week 2 | 447.6 (329.0)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 319.9 (453.8)
  Month 2: number analyzed (Participants) | 43
  Month 2 | 313.0 (707.9)
  Product Use End Visit: number analyzed (Participants) | 46
  Product Use End Visit | 296.6 (1099.2)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 2.8 (88.9)

19. Primary Outcome: Geometric Mean of Maternal TFV Concentrations From Breastmilk by Visit
Description: This endpoint is based on TFV concentration laboratory results from evaluable breastmilk specimens from mother participants. The geometric mean is summarized by study visit and includes only mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (1 ng/ml). The infant endpoints for geometric mean concentrations are included as separate sections below.
Time Frame: Measured through Month 3.5
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 48
ng/mL
  Week 1 | 5.6 (72.3)
  Week 2: number analyzed (Participants) | 47
  Week 2 | 4.3 (89.5)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 3.3 (108.3)
  Month 2: number analyzed (Participants) | 43
  Month 2 | 3.2 (120.0)
  Product Use End Visit: number analyzed (Participants) | 46
  Product Use End Visit | 2.7 (107.2)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 0.6 (106.5)

20. Primary Outcome: Geometric Mean of Infant DPV Concentrations From Plasma by Visit
Description: This endpoint is based on DPV concentration laboratory results from evaluable plasma specimens from infant participants. The geometric mean is summarized by study visit and includes only infants of mothers randomized to the DPV VR arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (20pg/ml). The mother endpoints for geometric mean concentrations are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Infants - Group A: DPV VR
Number analyzed (Participants) | 147
pg/mL
  Week 2: number analyzed (Participants) | 140
  Week 2 | 11.7 (46.3)
  Month 1: number analyzed (Participants) | 139
  Month 1 | 11.5 (35.7)
  Month 2: number analyzed (Participants) | 143
  Month 2 | 11.0 (31.7)
  Product Use End Visit: number analyzed (Participants) | 138
  Product Use End Visit | 10.5 (19.8)
  Study End Visit: number analyzed (Participants) | 142
  Study End Visit | 10 (0)

21. Primary Outcome: Geometric Mean of Infant FTC-TP Concentration by Visit
Description: This endpoint is based on FTC-TP concentration laboratory results from evaluable dried blood spot (DBS) specimens from infant participants. The geometric mean is summarized by study visit and includes only infants of mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (0.125 pmol/punch). The mother endpoints for geometric mean concentrations are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/punch
Arm/Group | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 48
pmol/punch
  Week 2: number analyzed (Participants) | 47
  Week 2 | 0.1 (23.5)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 0.1 (16.3)
  Month 2: number analyzed (Participants) | 45
  Month 2 | 0.1 (15.4)
  Product Use End Visit: number analyzed (Participants) | 45
  Product Use End Visit | 0.1 (12.1)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 0.1 (0)

22. Primary Outcome: Geometric Mean of Infant TFV-DP Concentrations by Visit
Description: This endpoint is based on TFV-DP concentration laboratory results from evaluable dried blood spot (DBS) specimens from infant participants. The geometric mean is summarized by study visit and includes only infants of mothers randomized to the Truvada arm. A value of 1/2 of the LLOQ is used if the concentration falls below the LLOQ (31.3 fmol/punch). The mother endpoints for geometric mean concentrations are included as separate sections above.
Time Frame: Measured through Month 3.5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/punch
Arm/Group | Infants - Group B: Truvada Tablet
Number analyzed (Participants) | 48
fmol/punch
  Week 2: number analyzed (Participants) | 47
  Week 2 | 15.6 (0)
  Month 1: number analyzed (Participants) | 47
  Month 1 | 15.6 (0)
  Month 2: number analyzed (Participants) | 45
  Month 2 | 15.6 (0)
  Product Use End Visit: number analyzed (Participants) | 45
  Product Use End Visit | 15.6 (0)
  Study End Visit: number analyzed (Participants) | 46
  Study End Visit | 15.6 (0)

23. Secondary Outcome: The Number of Mothers Non-adherent to Study Product for Each Month of Product Use by Study Product
Description: The number and proportion of mother's visits with drug concentration indicative of non-adherence (no use) are reported by study month. Non-adherence is measured by residual drug in returned VRs for mothers assigned the DPV VR arm and by TFV-DP concentrations in dried blood spot specimens for mothers assigned the Truvada tablet arm. For mothers on the DPV VR arm, no use is defined as residual DPV concentration in the returned VRs <= 0.9mg/month. For mothers on the Truvada arm, no use is defined as TFV-DP concentrations < 16.6 fmol/punch. Only mother participants are included in this endpoint since infants did not directly use study product in this study.
Time Frame: Measured through Month 3
Population: Only mother participants are included in this endpoint since infants did not directly use study product. The number of mothers analyzed includes mother participants with a returned/used vaginal ring that was successfully analyzed for residual drug concentration (evaluable) for Group A (DPV VR) and only those participants with an available and evaluable dried blood plot specimen for mothers in Group B (Truvada). Rings returned after the Month 3 Product Use End Visit (PUEV) are excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Non-adherence of Mothers randomized to the DPV VR study arm.
- Mothers - Group B: Truvada Tablet: Non-adherence of Mothers randomized to the Truvada oral tablet study arm.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 144 | 46
Participants
  Month 1: number analyzed (Participants) | 143 | 46
  Month 1 | 14 | 2
  Month 2: number analyzed (Participants) | 144 | 43
  Month 2 | 28 | 0
  Month 3: number analyzed (Participants) | 134 | 45
  Month 3 | 29 | 0

24. Secondary Outcome: Residual Drug Levels in Returned VRs
Description: The residual DPV concentrations from the returned VRs are summarized.
Time Frame: Measured through Month 3.5
Population: The analysis population includes mothers with evaluable residual DPV concentrations from returned vaginal rings (VRs). Rings returned on or after the Month 3 visit are included in the Month 3 summary.
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Mothers randomized to the DPV Vaginal Ring study arm with evaluable results for residual DPV concentrations from returned VRs.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004
Number analyzed (Participants) | 144
mg
  Month 1: number analyzed (Participants) | 143
  Month 1 | 22.1 [21.4 to 22.8]
  Month 2 | 22.4 [21.5 to 23.3]
  Month 3: number analyzed (Participants) | 137
  Month 3 | 22.1 [21.3 to 23.6]

25. Secondary Outcome: Participant Willingness to Use Their Assigned Study Products During Breastfeeding in the Future (Y/N)
Description: Based on participant report to the question "Would you be willing to use the study product for HIV prevention while breastfeeding in the future?"
Time Frame: Measured through Month 3.5
Population: The number of mothers analyzed includes all mothers who completed the Product End Use Visit Behavioral Assessment and responded to the willingness question. The count of participants who are willing, responded "Yes" to the question.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004: Mothers randomized to the Dapivirine (DPV) monthly Vaginal Ring (VR) study arm.
- Mothers - Group B: Truvada Tablet: Mothers randomized to the Truvada oral tablet study arm.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 145 | 48
Participants | 142 | 48

26. Secondary Outcome: Proportion of Participants Who Find Their Study Product to be at Least as Acceptable as Other HIV Prevention Methods
Description: Based on participant report on the question "Overall, how much did you like using the study product?" on the Product End Use Visit Behavioral Assessment.
Time Frame: Measured through Month 3.5
Population: The number of mothers analyzed included those who completed the Product End Use Visit Behavioral Assessment and responded to the acceptability question. The mothers who answered "Like very much" or "Like" are included in the total who find the study product acceptable.
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet
Number analyzed (Participants) | 145 | 47
Participants | 141 | 46

ADVERSE EVENTS:
Time Frame: The participant is followed for adverse events during study follow-up which was scheduled to be up to 14 weeks (98 days).
Description: The "Any Event in SOC" rows summarize the total number of adverse events within an SOC. In addition, these events are summarized using the specific Adverse Event Term for the event.
Arm/Group | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 | Mothers - Group B: Truvada Tablet | Infants - Group A: DPV VR | Infants - Group B: Truvada Tablet
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/49 | 0/148 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/148 | 0/49 | 4/148 | 0/49
Other Adverse Events (participants affected / at risk) | 92/148 | 35/49 | 112/148 | 32/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 (N=148) | Mothers - Group B: Truvada Tablet (N=49) | Infants - Group A: DPV VR (N=148) | Infants - Group B: Truvada Tablet (N=49)
Any Event in SOC (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers - Group A: Dapivirine (DPV) Vaginal Ring (VR)-004 (N=148) | Mothers - Group B: Truvada Tablet (N=49) | Infants - Group A: DPV VR (N=148) | Infants - Group B: Truvada Tablet (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micropenis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Eye disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 15 (16) | 11 (17) | 15 (16) | 5 (7)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 8 (8) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Any Event in SOC (General disorders) | 1 (1) | 3 (3) | 5 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Any Event in SOC (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess rupture (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 56 (73) | 17 (22) | 88 (179) | 26 (42)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 2 (2) | 5 (7) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 18 (18) | 6 (6)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 8 (9) | 5 (5) | 37 (56) | 11 (13)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (3)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea faciei (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 3 (3) | 40 (67) | 11 (15)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Vaccination site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 27 (31) | 17 (22) | 5 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 20 (20) | 13 (14) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 27 (34) | 10 (12)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 26 (33) | 10 (12)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 17 (20) | 2 (2) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Short stature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Any Event in SOC (Nervous system disorders) | 22 (28) | 8 (10) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (18) | 3 (3) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 14 (18) | 1 (1) | 0 (0) | 0 (0)
Cervix erythema (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Genital paraesthesia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 9 (9) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 24 (28) | 10 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (9) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04140266/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04140266/SAP_001.pdf